CLINICAL TRIAL: NCT00563498
Title: A Randomized Control Studies on the Effects of Glutamine on the Clinical Outcome of Bone Marrow Transplant Recipients With Special Reference to Veno-occlusive Disease and Mucositis.
Brief Title: Effects on Glutamine on the Outcome of Allogeneic Bone Marrow Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other); Fresienius Kabi HK Ltd (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC1432-00; HARECCTR0500034
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Pulmonary Veno-Occlusive Disease; Hepatic Veno-Occlusive Disease; Mucositis
Keywords: Veno-occlusive disease; Mucositis
MeSH Terms: conditions — Pulmonary Veno-Occlusive Disease; Hepatic Veno-Occlusive Disease; Mucositis | interventions — Glutamine

INTERVENTIONS:
Drug: Glutamine

SUMMARY:
The primary purpose of this project is to investigate if addition of glutamine, an amino acid, to standard parenteral nutrition, may improve the clinical outcome of the bone marrrow transplantation reducing the occurrence of veno-occlusive disease and severity of mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic bone marrow transplant recipients using busulfan and cyclophosphamide as conditioning.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-07; Study Completion 2006-06 (Estimated)

PRIMARY OUTCOMES:
Veno-occlusive disease | 1 month
Mucositis | 1 month

SECONDARY OUTCOMES:
Hospital stay | 2 months
Use of antibiotics | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lie, Dr, Principal Investigator — Department of Medicine/Division of Haematology, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China